CLINICAL TRIAL: NCT07338344
Title: Evaluation of the Clinical Efficacy and Safety of Luspatercept Combined With Low-dose Thalidomide Versus Luspatercept Alone in the Treatment of Adult Patients With Transfusion-dependent β-thalassemia
Brief Title: Evaluating the Clinical Efficacy and Safety of Luspatercept Combined With Thalidomide in the Treatment of β-TDT Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rongrong Liu (Other)
Responsible Party: Sponsor-Investigator, Rongrong Liu, consultant; professor, First Affiliated Hospital of Guangxi Medical University
Organization: First Affiliated Hospital of Guangxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-K0444
Record Dates: First submitted 2025-12-06; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Transfusion-dependent β-thalassemia Patients
MeSH Terms: interventions — Thalidomide; luspatercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial was conducted using a double-blind approach, meaning that neither the researchers nor the subjects knew the group assignments or the interventions they were receiving. Furthermore, the outcome assessors were also blinded, objectively evaluating the outcome measures without knowing the groups assigned to the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luspatercept(Reblozyl) combined with low-dose thalidomide (Experimental): The subjects in the intervention group were treated with Luspatercept (starting dose 1.0 mg/kg, once every 21 days) combined with low-dose thalidomide (starting dose level 50 mg/d) for 48 weeks.
  Interventions: Drug: Luspatercept combined with low-dose thalidomide
- Luspatercept plus placebo (Placebo Comparator): The control group was treated with Luspatercept (starting dose level 1.0 mg/kg every 21 days) plus placebo (starting dose level 50 mg/d) for 48 weeks.
  Interventions: Drug: Luspatercept plus placebo

INTERVENTIONS:
Drug: Luspatercept combined with low-dose thalidomide — The intervention group was treated with Luspatercept (starting dose level 1.0 mg/kg, once every 21 days) combined with low-dose thalidomide (starting dose level 50 mg/d) for 48 weeks.
  Arms: Luspatercept(Reblozyl) combined with low-dose thalidomide
Drug: Luspatercept plus placebo — The control group was treated with Luspatercept (starting dose level 1.0 mg/kg every 21 days) plus placebo (starting dose level 50 mg/d) for 48 weeks.
  Arms: Luspatercept plus placebo

SUMMARY:
β-thalassemia is one of the most common inherited hemoglobinopathies worldwide and a major public health issue that severely impacts birth quality, human health, and social progress. Currently, there are limited clinical drugs specifically designed to treat patients with β-thalassemia. This clinical trial aims to evaluate the efficacy and safety of luspatercept combined with low-dose thalidomide compared with luspatercept alone in patients with thalassemia. Key questions to be answered include:

* Does luspatercept combined with low-dose thalidomide reduce the transfusion burden in patients with β-thalassemia major?
* What medical problems may occur when patients receive luspatercept combined with low-dose thalidomide? In this clinical trial, participants were randomly assigned in a 1:1 ratio to either an intervention group (luspatercept combined with low-dose thalidomide) or a control group (luspatercept combined with placebo) using a central randomization system. The clinical efficacy and safety of the two groups were evaluated. The primary outcome measure was the clinical efficacy of luspatercept combined with low-dose thalidomide in reducing the transfusion burden in patients with β-thalassemia major.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the clinical efficacy and safety of luspatercept combined with low-dose thalidomide versus luspatercept combined with placebo in adult patients with β-thalassemia requiring regular red blood cell transfusions.

The study is divided into the following phases: screening/run-in period, double-blind treatment period, and follow-up period. Participants are centrally randomized in a 1:1 ratio to either the intervention group or the control group. The primary objective is to compare the clinical response rate between the intervention group (luspatercept combined with low-dose thalidomide) and the control group (luspatercept combined with placebo) in adult patients with transfusion-dependent β-thalassemia. Clinical response is defined as the proportion of subjects achieving a reduction in red blood cell (RBC) transfusion burden by ≥50% and at least 2 units during weeks 13-24 after randomization compared with the baseline period (12 weeks prior to randomization). Secondary objectives mainly include assessments of other clinical efficacy indicators, iron metabolism, hemolysis, as well as the incidence of adverse events.

Statistical analyses in this clinical study are based on the Intention-To-Treat (ITT) principle. Subgroup analyses of the primary endpoint are planned according to baseline transfusion burden (low, medium, and high transfusion burden groups).

The study plans to consecutively enroll 78 participants across eight research centers: the First Affiliated Hospital of Guangxi Medical University, Liuzhou People's Hospital, Liuzhou Worker's Hospital, Yulin First People's Hospital, Affiliated Hospital of Youjiang Medical University for Nationalities, Baise People's Hospital,Yunnan Provincial First People's Hospital and Southern Medical University Shenzhen Hospital. During the screening and run-in period, patients with severe β-thalassemia major (β-TM) who are scheduled to receive luspatercept combined with low-dose thalidomide or luspatercept monotherapy are invited to participate. Written informed consent is provided to potential subjects, along with a detailed explanation of the study content. Written informed consent from the subject (or their legal representative) must be obtained before any study-specific procedures are conducted. After signing the informed consent form, baseline data are collected. During the double-blind treatment period, the intervention group receives luspatercept combined with low-dose thalidomide, while the control group receives luspatercept combined with placebo. Both groups may receive best supportive care, including RBC transfusions, iron chelators, antiplatelet therapy, antibiotic therapy, antiviral and antifungal therapy, and/or nutritional support as needed. During the follow-up period, subjects are followed up at weeks 12, 24, 36, and 48. Data on physical examination, vital signs, hematological tests, clinical biochemistry, transfusion status, iron parameters, quality of life, concomitant treatments, subject compliance, and adverse events are collected and recorded in detail for further analysis of clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, regardless of gender;
* Patients with transfusion-dependent β-thalassemia;
* Intended treatment with rotecept combined with low-dose thalidomide or rotecept alone;
* Requires regular red blood cell transfusions (6-30 RBC units (International Units) within 24 weeks prior to randomization, with a transfusion-free interval of ≤ 42 days);
* ECOG performance status 0-1;
* Patients (or legal guardians) voluntarily participate in the study and provide signed informed consent.

Exclusion Criteria:

* A diagnosis of α-thalassemia minor, Hb Bart's edema, hemoglobin S/β-thalassemia, or myelodysplastic anemia (combination of β-thalassemia and α-thalassemia is permitted);
* Anemia related to nutritional deficiency, anemia of chronic disease, autoimmune hemolytic anemia, or any other hemolytic anemia (e.g., severe G6PD deficiency, pyruvate kinase deficiency);
* A bleeding disorder manifesting as frequent bleeding (e.g., menorrhagia, epistaxis, coagulopathy);
* Hemolysis unrelated to thalassemia within the past 8 weeks, such as after use of hemolytic-inducing medications (e.g., antimalarials, nonsteroidal anti-inflammatory drugs [NSAIDs]);
* Use of long-term anticoagulant therapy, unless discontinued at least 28 days before randomization. Prophylactic anticoagulant therapy for surgery or high-risk procedures, as well as low-molecular-weight heparin and long-term aspirin therapy for superficial venous thrombosis, are permitted.
* Use of thalidomide alone, erythropoiesis-stimulating drugs (ESA), or hydroxyurea within the past 24 weeks.
* Use of long-term systemic glucocorticoids within the past 12 weeks.
* Use of cytotoxic drugs, immunosuppressants, or other investigational drugs within the past 28 days.
* HIV positive and/or active HCV or HBV infection.
* Hepatic and renal insufficiency (liver insufficiency, i.e., aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≥3× upper limit of normal (ULN); renal insufficiency, i.e., serum creatinine ≥3× upper limit of normal (ULN) or creatinine clearance less than 30). mL/min), history of malignancy (unless cured and/or with no known active disease);
* Women who are pregnant, plan to become pregnant during the study, or are breastfeeding;
* Previous thalassemia gene therapy or hematopoietic stem cell transplantation (HSCT);
* Platelet count < 70 × 109/L, if not associated with hypersplenism, or platelet count > 1,000 × 109/L;
* Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved Erythroid Response - Week 13 to Week 24 | Baseline: Day -83 to Day 1; Treatment: Weeks 13 to Week 24
  Percentage of participants with a ≥50% reduction in RBC transfusion burden compared to baseline (RBC transfusion burden during the 12 weeks before randomization) and a reduction of at least 2 units for 12 consecutive weeks between Weeks 13 and 24 after randomization

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved ≥ 50% And a Reduction of ≥ 2 RBC units From Baseline in Transfusion Burden- Week 37 to Week 48 | Baseline: Day -83 to Day 1; Treatment: Weeks 37 to Week 48
  Percentage of participants who achieved a ≥50% reduction in RBC transfusion burden relative to baseline, with a reduction of ≥ 2 RBC units, for 12 consecutive weeks between 37 and 48 weeks after randomization.
Percentage Of Participants Who Achieved ≥ 33% And a Reduction of ≥ 2 RBC units Reduction From Baseline in Transfusion Burden - Week 37 to Week 48 | Baseline: Day -83 to Day 1; Treatment: Weeks 37 to Week 48
  Percentage Of participants who achieved a ≥33% reduction in RBC transfusion burden relative to baseline, with a reduction of ≥ 2 RBC units, for 12 consecutive weeks between 37 and 48 weeks after randomization.
Percentage Of Participants Who Achieved ≥ 50% Reduction From Baseline in Transfusion Burden - weeks 1-12, 13-24, 25-36, 37-48 | Baseline: Day -83 to Day 1; Treatment: Weeks1-12, 13-24, 25-36, 37-48
  Percentage Of participants who achieved a ≥50% reduction in RBC transfusion burden relative to baseline (RBC transfusion burden during the 12 weeks prior to randomization) for any consecutive 12 weeks (weeks 1-12, 13-24, 25-36, 37-48).
Percentage Of Participants Who Achieved ≥ 33% Reduction From Baseline in Transfusion Burden - weeks 1-12, 13-24, 25-36, 37-48 | Baseline: Day -83 to Day 1; Treatment: Weeks1-12, 13-24, 25-36, 37-48
  Percentage Of participants who achieved a ≥33% reduction in RBC transfusion burden relative to baseline (RBC transfusion burden during the 12 weeks prior to randomization) for any consecutive 12 weeks (weeks 1-12, 13-24, 25-36, 37-48).
Percentage Of Participants Who Achieved ≥ 50% Reduction From Baseline in Transfusion Burden - weeks 1-24, 25-48 | Baseline: Day -83 to Day 1; Treatment: Weeks1-24, 25-48
  Percentage Of participants with a ≥50% reduction in RBC transfusion burden relative to baseline (RBC transfusion burden during the 12 weeks prior to randomization) during any 24 consecutive weeks (weeks 1-24, 25-48);
Percentage Of Participants Who Achieved ≥ 33% Reduction From Baseline in Transfusion Burden - weeks 1-24, 25-48 | Baseline: Day -83 to Day 1; Treatment: Weeks1-24, 25-48
  Percentage Of participants with a ≥33% reduction in RBC transfusion burden relative to baseline (RBC transfusion burden during the 12 weeks prior to randomization) during any 24 consecutive weeks (weeks 1-24, 25-48);
Maximum percentage change in transfusion burden from baseline over 12 consecutive weeks | Baseline: Day -83 to Day 1; Treatment: Weeks1-12, 13-24, 25-36, 37-48
  Percentage Of participants change in RBC transfusion burden relative to baseline (RBC transfusion burden during the 12 weeks prior to randomization) during any 12 consecutive weeks (weeks 1-12, 13-24, 25-36, 37-48);
Percentage of Participants Who Maintained Red Blood Cell (RBC) Transfusion Independence For ≥8 Weeks | weeks 1-8, 9-16, 17-24, 25-32, 33-40, 41-48
  Percentage of Participants who became transfusion-independent during any 8 consecutive weeks (weeks 1-8, 9-16, 17-24, 25-32, 33-40, 41-48);
Percentage of Participants Who Maintained Red Blood Cell (RBC) Transfusion Independence For ≥12 Weeks | weeks 1-12, 13-24, 25-36, and 37-48
  Percentage of Participants who became transfusion-independent during any 12 consecutive weeks (weeks 1-12, 13-24, 25-36, and 37-48);
Maximum percentage change from baseline in the number of transfusion events over 12 consecutive weeks | Baseline: Day -83 to Day 1; Treatment: Weeks1-12, 13-24, 25-36, 37-48
  Maximum percentage change from baseline in the number of transfusion events (RBC transfusion burden during the 12 weeks prior to randomization) during any 12 consecutive weeks (weeks 1-12, 13-24, 25-36, and 37-48);
Concentration Change From Baseline to End of Treatment in serum ferritin | Baseline (prior to first dose of study drug) and Treatment (weeks 12,24,36,48)
  Concentration change from baseline in serum ferritin at weeks 12, 24, 36, and 48 after randomization;
Change From Baseline to End of Treatment in Iron deposition in organs | Baseline (prior to first dose of study drug) and Treatment (weeks 24,48)
  Change from baseline in myocardial iron and liver iron concentrations at weeks 24 and 48 after randomization;
Change From Baseline to End of Treatment in the average daily dose of iron chelation therapy | Baseline (prior to first dose of study drug) and Treatment (weeks 1-48)
  Change from baseline in the average daily dose of iron chelation therapy (ICT) during the treatment period (up to 48 weeks);
Change from baseline in self-reported Health-related quality-of-life (HRQoL) assessed by TranQoL | Baseline (prior to first dose of study drug) and Treatment (weeks 24,48)
  The TranQol is a self-administered quality of life tool developed for beta-thalassemia patients. The adult self-report version used in this study, includes 36 questions assessed on a 5-point response, that are grouped into 5 domains (Physical Health, Emotional Health, Sexual Health, Family Functioning, School/Career Functioning). Scores are calculated according to specific scoring algorithms developed by the authors. Both individual domains score and the total score range from 0 (worst) to 100 (best). Total Score and Physical Health domain score are reported. Positive change from baseline values indicate improvement.
Change from baseline in self-reported Health-related quality-of-life (HRQoL) assessed by SF-36 | Baseline (prior to first dose of study drug) and Treatment (weeks 24,48)
  The SF-36 (version 2) is a generic, self-administered instrument consisting of 8 multi-item scales that assess 8 health domains. The raw score for each health domain is transformed into a 0 (worst) to 100 (best) domain score. The 0-100 scale score for each health domain is further converted to normbased scores using a T-score transformation, with a mean of 50 and a standard deviation (SD) of 10. Higher norm-based T-scores indicate better heath/QoL. The domains/summaries reported are: 1. Physical Functioning (Range of possible T-scores is 19.26 - 57.54) 2. General Health (Range of possible T-scores is 18.95 - 66.50) 3. Physical Component summary (PCS) (Range of possible T-scores is 5.02 - 79.78). Positive change from baseline values indicate improvement.

OTHER OUTCOMES:
Percent Change From Baseline to End of Treatment in Fetal hemoglobin | Baseline (prior to first dose of study drug) and Treatment (weeks 12,24,36,48)
  Percent changes from baseline in fetal hemoglobin (HbF) at weeks 12, 24, 36, and 48 after randomization
Change From Baseline to End of Treatment in γ-Globin Gene | Baseline (prior to first dose of study drug) and Treatment (weeks 12,24,36,48)
  Change from baseline to end of treatment in γ-globin geneγ-globin gene expression at weeks 12, 24, 36, and 48 after randomizatio
Concentration Change From Baseline to End of Treatment in Hemolysis Indices | Baseline (prior to first dose of study drug) and Treatment (weeks 12,24,36,48)
  Changes in concentration values from baseline to end of treatment in hemolysis indices the changes in hemolysis indicators (total bilirubin (TIBL), indirect bilirubin (IBIL), lactate dehydrogenase (LDH), and reticulocytes) relative to baseline at weeks 12, 24, 36, and 48 after randomization
Safety - Incidence of Adverse Events (AEs) | Weeks1--48
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. A serious AE is any AE occurring at any dose that - Results in death - Is life-threatening - Requires or prolongs existing inpatient hospitalization - Results in persistent or significant disability/incapacity - Is a congenital anomaly/birth defect - Constitutes an important medical event. The Investigator assessed the relationship of each AE to study drug and graded the severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03): - Grade 1 = Mild - Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention) - Grade 3 = Severe (limitation in activity; medical intervention required) - Grade 4 = Life-threatening - Grade 5 = Death.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Southern Medical University Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Youjiang Medical College for Nationalities, Baise City, Guangxi
  - Baise People's Hospital, Baise City, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - Yulin First People's Hospital, Yulin, Guangxi
  - Yunnan Provincial First People's Hospital, Kunming, Yunnan
  - The First Affiliated Hospital of Guangxi Medical University, Naning

IPD SHARING:
Plan to Share IPD: No